CLINICAL TRIAL: NCT06213675
Title: A Randomized Controlled Study to Explore the Effect of Intra-articular Injection on Temporomandibular Joint Dysfunction
Brief Title: Effect of Intra-articular Injection on Temporomandibular Joint Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KY-0107-011
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Temporomandibular Joint Dysfunction
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Injections, Intra-Articular

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental): The patients receive a 15-day treatment and are required to stay in the hospital during this period. Patients in the experimental group are given routine rehabilitation treatment and intra-articular injections. Lidocaine is used as the injected medication at a dose of 2ml, administered once every 5 days for a total of three injections.
  Interventions: Behavioral: Routine rehabilitation treatment; Procedure: Intra-articular Injection
- The control group (Active Comparator): The patients receive a 15-day treatment and are required to stay in the hospital during this period. Patients are given routine rehabilitation treatment.
  Interventions: Behavioral: Routine rehabilitation treatment

INTERVENTIONS:
Behavioral: Routine rehabilitation treatment — Routine rehabilitation treatment Includes oral rehabilitation, rehabilitation training for temporomandibular disorders, orthodontic treatment, and other physical therapy methods.which can alleviate symptoms by adjusting the bite, relaxing muscles, and increasing the range of motion of the temporomandibular joint.
  Besides, it also Includes temporomandibular joint exercise training, relaxation training for facial muscles, and functional chewing training aimed at improving temporomandibular joint function and muscle balance.
Procedure: Intra-articular Injection — The patient is positioned to maximize mouth opening, and a needle is inserted approximately 10-12 mm in front of the tragus after touching the ankle prominence. An 8# injection needle is chosen and inserted upward and slightly forward into the joint cavity. A total of 2 mL of lidocaine hydrochloride injection solution is injected, repeated once every 5 days for a total of 15 days.
  Arms: the experimental group

SUMMARY:
The goal of this clinical trial is to study about the clinical effect of Intra-articular Injection on Temporomandibular Joint Dysfunction

The main question it aims to answer is:

• Can Intra-articular Injection help improve the Temporomandibular Joint Dysfunction Participants will be randomly assigned into the experimental group and the control group, all under comprehensive treatment. The experimental group will be given Intra-articular Injection additionally, The study lasts 15 days for each patient. Researchers will compare the assessments between the two groups to see if Intra-articular Injection can help improve the Temporomandibular Joint Dysfunction

DETAILED DESCRIPTION:
The background of Temporomandibular Joint Dysfunction is that it is one of the common diseases in the oral and maxillofacial region, and it is the most common among temporomandibular joint diseases. It is more prevalent in young adults, with the highest prevalence rate at 20-30 years old.

The goal of this clinical trial is to study about the clinical effect of Intra-articular Injection on Temporomandibular Joint Dysfunction

The main question it aims to answer is:

• Can Intra-articular Injection help improve the Temporomandibular Joint Dysfunction Participants will be randomly assigned into the experimental group and the control group, all under comprehensive treatment. The experimental group will be given Intra-articular Injection additionally, The study lasts 15 days for each patient. Researchers will compare the assessments between the two groups to see if Intra-articular Injection can help improve the Temporomandibular Joint Dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Presence of significant temporomandibular disorder clinical symptoms.
* Meeting the diagnostic criteria for Temporomandibular Joint Dysfunction and confirmed by X-ray examination.
* Patients voluntarily participate in this study and provide signed informed consent.
* Normal cognitive function

Exclusion Criteria:

* Rheumatic, rheumatoid, or other severe systemic diseases.
* Infectious temporomandibular joint arthritis or joint tumors.
* Individuals who have recently received joint injection treatment or photodynamic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Friction Index | day 1 and day 15
  Friction Index is used to assess temporomandibular function. The total scores range from 0 to 57, with higher scores indicating more severe temporomandibular dysfunction.

SECONDARY OUTCOMES:
The Visual Analog Scale | day 1 and day 15
  The Visual Analog Scale is used to assess the pain levels of two groups of patients. The total score ranges from 0 to 10, with higher scores indicating more severe pain.
The maximum mouth opening limit | day 1 and day 15
  The maximum mouth opening limit is measured with precision to 0.1 mm (the distance between the upper and lower lips).
Mann Assessment of Swallowing Ability | day 1 and day 15
  Mann Assessment of Swallowing Ability is used to assess swallowing function. The maximum score on the scale is 200. Each item on the scale is scored from 0 to 6, and the total score is calculated by summing up the scores across all items. A higher score indicates better swallowing ability, while a lower score suggests the presence of swallowing difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Zheng Da yi Yuan Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No